CLINICAL TRIAL: NCT00745212
Title: Prospective Multicentric Evaluation of an Antithrombotic Therapeutic Strategy in Pregnant Women With a Risk of Thromboembolism and/or a Risk of Placental Vascular Complication, Strategy Determined With a Risk Score.
Brief Title: Evaluation of an Antithrombotic Therapeutic Strategy in Pregnant Women
Acronym: STRATHEGE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0508080
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Placental Vascular Pathologies; Venous Thromboembolism Diseases
Keywords: venous thromboembolism diseases; placental vascular pathologies; antithrombotic treatment; symptomatic thromboembolic events; pregnant women; score; therapeutic strategies; heparin; aspirin; pregnancy pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The venous thromboembolism is one of the first causes of maternal mortality. Until 2003, only a few recommendations were available on the optimal use of antithrombotic therapy as a preventive measure against thromboembolism in pregnant women. In this study, we propose :

1. To gather the experts who took part in the French consensus conference and the local experts to create a score in accordance with the national and international consensus and to give some precise therapeutic strategies.
2. To evaluate the discriminant, feasible and useful character of this new score by a prospective multicentric study including 2000 pregnant women with a risk of thromboembolism or placental vascular pathology who will benefit from therapeutic strategies defined by the new score.

   .

DETAILED DESCRIPTION:
Purpose : To create a score inspired by our first experience i.e. simple, standardized and quickly usable in day-to-day practice to individualize antithrombotics prescription to women at risk.

ELIGIBILITY:
Inclusion Criteria:

* multiparous or primiparous parturients followed in one of the participating centers
* Presenting at least one risk factor of venous thromboembolic pathology and/or placental vascular pathology

Exclusion Criteria:

* parturient that can't be followed
* unknown familial or personal previous history
* Parturient with a contraindication to use of the treatment recommended by the therapeutic strategy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 2280 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Occuring of symptomatic thromboembolic events and/or placental vascular pathology, any other pregnancy pathology requiring hospitalization, any complications from the antithrombotic treatment | first, second or third trimester during pregnancy or post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Céline CHAULEUR, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Service de Gynécologie Obstétrique - CHU Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Derived] Chauleur C, Gris JC, Laporte S, Rancon F, Varlet MN, Decousus H, Mismetti P; STRATHEGE Group. Use of the Delphi method to facilitate antithrombotics prescription during pregnancy. Thromb Res. 2010 Aug;126(2):88-92. doi: 10.1016/j.thromres.2010.01.012. Epub 2010 Feb 13. PMID 20153880